CLINICAL TRIAL: NCT00747851
Title: NETs: Protection or Harm in Neonatal Inflammation or Infection
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christian Con Yost, Principal Investigator, University of Utah
Other Study IDs: 11919; R01HD093826 (NIH)
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Necrotizing Enterocolitis (NEC)
Keywords: protein; synthesis; response; PAF-stimulated; PMNs; collected
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective in vitro cell biology study of polymorphonuclear leukocyte (PMN) protein synthesis in response to PAF. PMNs from cord blood of premature human infants at risk for NEC (birth weight between 501 - 1500 grams) and PMNs from cord blood of healthy term infants will be isolated and stimulated with PAF, a biologically active phospholipid implicated in the pathogenesis of NEC. NEC, a disease of prematurity with an incidence of 10.1% of infants born weighing between 501 - 1500 grams, is associated with significant morbidity and mortality. We will compare the protein synthesis of inflammatory modulators, including Interleukin 6 Receptor alpha (IL-6R alpha) and Retinoic Acid Receptor alpha (RAR alpha) proteins to protein synthesis responses already observed in PMNs isolated from healthy adults. Furthermore, we will characterize the expression and activity of the mammalian target of rapamycin (mTOR) translational protein synthesis control pathway in PMNs isolated from preterm and term infants and compare those results with previous observations in PMNs isolated from adults. This pathway is known to regulate IL-6R alpha and RAR alpha protein expression in PMNs isolated from adults. We will also follow those premature infants at risk for NEC clinically to determine which infants develop NEC and what risk factors may be associated with NEC in this population.

DETAILED DESCRIPTION:
Many pediatric diseases including Systemic Inflammatory Response Syndrome (SIRS), sepsis, Acute Respiratory Distress Syndrome (ARDS) and neonatal Chronic Lung Disease (CLD) have been associated with dysregulation of the acute inflammatory response [1]. So it is with necrotizing enterocolitis (NEC). NEC, a disease of premature infants, afflicts 10% of very low birth weight infants. This disease is often fatal [2]. Less significant but nonetheless devastating sequelae include intestinal perforation, short gut syndrome, prolonged total parenteral nutrition with possible concomitant liver failure and a prolonged intensive care unit stay. The etiology remains unknown, although risk factors of prematurity, enteral feeds, infection and intestinal ischemia are associated with NEC [3].

The final common pathway for NEC appears, at least in part, to be mediated through the biologically active phospholipid platelet-activating factor (PAF). Each identified risk factor for NEC increases the serum levels of PAF in premature infants[4, 5]. Furthermore, serum levels of PAF-acetylhydrolase (PAF-AH), the enzyme responsible for catabolizing PAF, are lower in premature infants compared to term infants and lower in term infants compared to young children and adults [6, 7]. Although no clinical trials of PAF antagonists have been conducted in premature human infants, various PAF antagonists prevent NEC-like clinical disease in animal models [8-10].

Other data from animal models suggest a prominent role of the polymorphonuclear leukocyte (PMN) in the pathogenesis of NEC. Musemeche et al. induced NEC-like disease in rats by intra-aortic injection of PAF [11]. They used vinblastine, a chemotherapeutic agent with a side-effect profile significant for induction of neutropenia, to induce neutropenia in rats four days prior to intra-aortic injection of PAF. The vinblastine-induced neutropenia was protective for the clinical and pathologic manifestations of NEC-like disease. Other investigators have demonstrated an increase in PAF levels in the gastrointestinal tracts of rats subjected to gut ischemia/reperfusion. The elevated levels of intestinal PAF were then shown to chemo attract and prime PMNs [12].

The role of the human PMN in the acute inflammatory response is well documented. They play a fundamental role in the non-specific immune response and are rapidly recruited to areas of injury or inflammation where they participate in bacterial phagocytosis and killing. Disorders associated with a deficiency or impairment of PMNs (neutropenia, chronic granulomatous disease, leukocyte adhesion deficiency) predispose to infections with gram-negative and gram-positive bacteria [13]. However, regulation of this potent component of the acute inflammatory response is imperative. Disorders such as ARDS, ischemia/reperfusion injury and rheumatoid arthritis appear to result from the dysregulation of the PMNs' acute inflammatory response [1].

The molecular mechanisms regulating the PMNs' response in acute inflammation are not fully understood. In neutrophil priming, the activation of the NADPH oxidase enzyme via receptor-mediated stimulation with mediators such as fMLP or PAF is an increasingly complex process involving various cellular secondary messengers and the Rho family GTPase Rac2 [14, 15]. The mechanisms regulating PMN synthesis and release of pro-inflammatory cytokines such as IL-8 are less well understood. The mechanisms regulating PMN apoptosis are also not well understood. In vitro and in vivo studies indicate that the pro-inflammatory agents responsible for the priming of human PMNs also affect the longevity of those cells by delaying the PMNs in-built capacity to undergo apoptosis. In vitro studies on human PMNs show that pro-inflammatory mediators like Granulocyte/Macrophage - Colony Stimulating Factor (GM-CSF), Interleukin-8 (IL-8), Lipopolysaccharide (LPS), Complement 5a (C5a) and Interleukin-6 (IL-6) inhibit PMN apoptosis, while Tumor Necrosis Factor (TNF) and Fas-ligand (Fas-L) accelerate the rate of neutrophil apoptosis [16].

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the NICU who were less than or equal to 1500 grams or less than 30 weeks gestational age at birth; Term infants delivered at UUMC without complication, either via cesarean section or vaginal delivery; Cord blood isolated within first hour of life; and parents or guardians must have signed informed consent.

Exclusion Criteria:

* Infants with major congenital anomalies will be excluded.

Max Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients hospitalized in the NICU who were less than or equal to 1500 grams or less than 30 weeks gestational age at birth
Sampling Method: Non-Probability Sample
Enrollment: 388 (Estimated)
Dates: Start 2003-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and survival of premature infants with NEC, defined prospectively as disease meeting criteria for Bell's classification category IIA or greater [See Table 1] as applied by the subject's attending physician. | 2 years

SECONDARY OUTCOMES:
Multiple morbidities and other clinical data will be collected and evaluated with respect to NEC and PMN protein analysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Yost, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States